CLINICAL TRIAL: NCT04949620
Title: REThinkWELL: An Evidence-based Integrative Platform for the Prevention of Emotional Disorders in Children and Promotion of Children's Emotional Health
Brief Title: An Integrative Platform for Promoting Children's Emotional Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Collaborators: The Executive Agency for Higher Education, Research, Development and Innovation Funding (Other)
Responsible Party: Principal Investigator, Oana David, Professor, Babes-Bolyai University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 2576/ 18.03.2021
Record Dates: First submitted 2021-05-11; First posted 2021-07-02 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Emotional Problem
Keywords: emotional problems; children; parenting; online therapeutic game

STUDY DESIGN:
Intervention Model Description: The first stage investigates the efficacy of the online REThink therapeutic game in comparison with monitoring in the prevention of emotional disorders for 4 weeks. In the second stage, for the non-responders to the intervention, the online parenting intervention will be implemented, while the other groups will be monitored for other 4 weeks.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- REThink game, then responder monitoring (Experimental): Participants in this group will have access to the REThink game for four weeks; based on their response to the intervention, they will be monitored for an additional period of four weeks.
  Interventions: Behavioral: REThink therapeutic game
- REThink game, then online parent intervention for non-responders (Experimental): Participants who are allocated to the REThink game and do not respond to the four-week intervention will be allocated to the online
  Interventions: Behavioral: REThink therapeutic game; Behavioral: Online parenting program
- Monitoring (No Intervention): Participants in this arm will be monitored for a total of eight weeks, for comparison with the REThink game intervention (after four weeks) and the online parenting program (after an additional four weeks).

INTERVENTIONS:
Behavioral: REThink therapeutic game — REThink is a online therapeutic game developed by David and collaborators (2018), proved to be an efficient intervention for the reduction of emotional symptoms in children and adolescents.
  Arms: REThink game, then online parent intervention for non-responders; REThink game, then responder monitoring
Behavioral: Online parenting program — The online parenting intervention consists of a newly developed parenting program, including rational emotive behavioral therapy and schema therapy principles
  Arms: REThink game, then online parent intervention for non-responders

SUMMARY:
The general objective of the study is to test an online platform for the promotion of emotional health in children

DETAILED DESCRIPTION:
The project aims at implementing an integrated online therapeutic platform that will be accessed by youth, parents and clinicians. The main original feature is the integration of state of the art online/mobile and gaming technologies into a unique platform that allows easy access to personalized, accessible and validated prevention.

The platform aims to allow access to attractive, easily accessible and evidence-based prevention for youths. The system will be validated in the second step as an integrative, multi-componential and adaptive platform for the prevention of emotional disorders in youth. The platform includes tools that were separately tested in laboratory conditions and found to be effective: the REThink therapeutic video game and the online REThink Parenting and Rational Parent Coach mobile programs.

ELIGIBILITY:
Inclusion Criteria:

* children aged 8 to 12 years
* scores above average at any subscale of Childhood Trauma Questionnaire
* parental consent provided
* for the parental intervention: no changes in children's main outcomes following the REThink intervention

Exclusion Criteria:

* intellectual disability or physical limitations precluding the use of the online platform
* presence of a mental health disorder in the children or their enrolled parent

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 256 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Children's emotional symptoms | baseline
  The Child Behavior Checklist for ages 6-18 (CBCL; Achenbach & Rescorla, 2001) is a parent-report of child emotional and behavioral problems. Each item is rated on a 3-point Likert-style scale ranging from 0 (not true) to 2 (very true or often true). The DSM-derived affective and anxiety scales and the anxious/depressed and withdrawn/depressed syndrome scales, respectively, will be used to assess emotional symptoms.
Changes in children's emotional symptoms - immediately | immediately post first-stage intervention (4 weeks following baseline)
  The Child Behavior Checklist for ages 6-18 (CBCL; Achenbach & Rescorla, 2001) is a parent-report of child emotional and behavioral problems. Each item is rated on a 3-point Likert-style scale ranging from 0 (not true) to 2 (very true or often true). The DSM-derived affective and anxiety scales and the anxious/depressed and withdrawn/depressed syndrome scales, respectively, will be used to assess emotional symptoms.

SECONDARY OUTCOMES:
Child irrationality | baseline
  The Child and Adolescent Scale of Irrationality "Bernard ME, Cronan F (1999) The child and adolescent scale of irrationality: validation data and mental health correlates. J Cogn Psychother 13:121-132"
Child trauma | baseline
  CTQ - Childhood Trauma Questionnaire Bernstein, D. P., Stein, J. A., Newcomb, M. D., Walker, E., Pogge, D., Ahluvalia, T., ... & Zule, W. (2003). Development and validation of a brief screening version of the Childhood Trauma Questionnaire. Child abuse & neglect, 27(2), 169-190.
Child behavioral difficulties | baseline
  SDQ - Strengths and Difficulties Questionnaire "Goodman R, Meltzer H, Bailey V (1998) The strengths and difficulties questionnaire: "a pilot study on the validity of the self-report version. Eur Child Adolesc Psychiatry 7:125-130"
Changes in child irrationality | immediately post first-stage intervention (4 weeks following baseline)
  The Child and Adolescent Scale of Irrationality "Bernard ME, Cronan F (1999) The child and adolescent scale of irrationality: validation data and mental health correlates. J Cogn Psychother 13:121-132"
Changes in child behavioral difficulties | immediately post first-stage intervention (4 weeks following baseline)
  SDQ - Strengths and Difficulties Questionnaire "Goodman R, Meltzer H, Bailey V (1998) The strengths and difficulties questionnaire: "a pilot study on the validity of the self-report version. Eur Child Adolesc Psychiatry 7:125-130"
Changes in children emotional abilities | immediately post first-stage intervention (4 weeks following baseline)
  The Cognitive Emotion Regulation Questionnaire - Short (Garnefski & Kraaij, 2006) is an 18-item self-report scale that measures a total of nine different cognitive coping strategies, each addressed by two items.

OTHER OUTCOMES:
Parenting practices | immediately post first-stage intervention (4 weeks following baseline)
  The Parenting to Reduce Adolescent Depression and Anxiety Scale (PRADAS; Cardamone-Breene et al., 2017) is a 79-item self-report measure of parenting practices. The instrument comprises nine subscales (6-12 items each), corresponding to nine sets of parenting practices that are part of the national Australian guidelines for helping reduce depression in children and adolescents. Most items are scored on a Likert scale measuring the frequency of distinct parenting behaviors (never, rarely, sometimes, and often).
Changes in parenting practices | post second-stage intervention (8 weeks following baseline)
  The Parenting to Reduce Adolescent Depression and Anxiety Scale (PRADAS; Cardamone-Breene et al., 2017) is a 79-item self-report measure of parenting practices. The instrument comprises nine subscales (6-12 items each), corresponding to nine sets of parenting practices that are part of the national Australian guidelines for helping reduce depression in children and adolescents. Most items are scored on a Likert scale measuring the frequency of distinct parenting behaviors (never, rarely, sometimes, and often).
Changes in parenting practices - follow up | 6-month follow-up
  The Parenting to Reduce Adolescent Depression and Anxiety Scale (PRADAS; Cardamone-Breene et al., 2017) is a 79-item self-report measure of parenting practices. The instrument comprises nine subscales (6-12 items each), corresponding to nine sets of parenting practices that are part of the national Australian guidelines for helping reduce depression in children and adolescents. Most items are scored on a Likert scale measuring the frequency of distinct parenting behaviors (never, rarely, sometimes, and often).
Changes in parenting practices - follow up one year | 12-month follow-up
  The Parenting to Reduce Adolescent Depression and Anxiety Scale (PRADAS; Cardamone-Breene et al., 2017) is a 79-item self-report measure of parenting practices. The instrument comprises nine subscales (6-12 items each), corresponding to nine sets of parenting practices that are part of the national Australian guidelines for helping reduce depression in children and adolescents. Most items are scored on a Likert scale measuring the frequency of distinct parenting behaviors (never, rarely, sometimes, and often).
Parent distress | immediately post first-stage intervention (4 weeks following baseline)
  The Profile of Emotional Distress (PED; Opris & Macavei, 2005) is a is a 40-item self-report instrument measuring functional and dysfunctional negative emotions based on Albert Ellis's binary model of distress, as well as positive emotions. The negative emotion subscales include two dysfunctional emotion dimensions (anxiety and depression) and two functional counterparts (concern and sadness). Responders are asked to assess the degree to which they have experienced each emotion during the previous two weeks, based on a five-point Likert scale ranging from "Not at all" (0) to "Extremely" (4).
Changes in parent distress | post second-stage intervention (8 weeks following baseline)
  The Profile of Emotional Distress (PED; Opris & Macavei, 2005) is a is a 40-item self-report instrument measuring functional and dysfunctional negative emotions based on Albert Ellis's binary model of distress, as well as positive emotions. The negative emotion subscales include two dysfunctional emotion dimensions (anxiety and depression) and two functional counterparts (concern and sadness). Responders are asked to assess the degree to which they have experienced each emotion during the previous two weeks, based on a five-point Likert scale ranging from "Not at all" (0) to "Extremely" (4).
Changes in parent distress -follow up | 6-month follow-up
  The Profile of Emotional Distress (PED; Opris & Macavei, 2005) is a is a 40-item self-report instrument measuring functional and dysfunctional negative emotions based on Albert Ellis's binary model of distress, as well as positive emotions. The negative emotion subscales include two dysfunctional emotion dimensions (anxiety and depression) and two functional counterparts (concern and sadness). Responders are asked to assess the degree to which they have experienced each emotion during the previous two weeks, based on a five-point Likert scale ranging from "Not at all" (0) to "Extremely" (4).
Changes in parent distress -follow up one year | 12-month follow-up
  The Profile of Emotional Distress (PED; Opris & Macavei, 2005) is a is a 40-item self-report instrument measuring functional and dysfunctional negative emotions based on Albert Ellis's binary model of distress, as well as positive emotions. The negative emotion subscales include two dysfunctional emotion dimensions (anxiety and depression) and two functional counterparts (concern and sadness). Responders are asked to assess the degree to which they have experienced each emotion during the previous two weeks, based on a five-point Likert scale ranging from "Not at all" (0) to "Extremely" (4).
Parent beliefs | immediately post first-stage intervention (4 weeks following baseline)
  The Parent Rational and Irrational Beliefs Scale (P-RIBS; Gavita, DiGiuseppe, David & DelVecchio, 2011) is a 24-item measure of rational and irrational evaluative processes in parents regarding child behavior and the parent role. Items are assessed on a 5- point Likert scale, from "Strongly disagree" (1) to "Strongly agree" (5).
Changes in parent beliefs | post second-stage intervention (8 weeks following baseline)
  The Parent Rational and Irrational Beliefs Scale (P-RIBS; Gavita, DiGiuseppe, David & DelVecchio, 2011) is a 24-item measure of rational and irrational evaluative processes in parents regarding child behavior and the parent role. Items are assessed on a 5- point Likert scale, from "Strongly disagree" (1) to "Strongly agree" (5).
Changes in parent beliefs - follow up | 6-month follow-up
  The Parent Rational and Irrational Beliefs Scale (P-RIBS; Gavita, DiGiuseppe, David & DelVecchio, 2011) is a 24-item measure of rational and irrational evaluative processes in parents regarding child behavior and the parent role. Items are assessed on a 5- point Likert scale, from "Strongly disagree" (1) to "Strongly agree" (5).
Changes in parent beliefs - follow up one year | 12-month follow-up
  The Parent Rational and Irrational Beliefs Scale (P-RIBS; Gavita, DiGiuseppe, David & DelVecchio, 2011) is a 24-item measure of rational and irrational evaluative processes in parents regarding child behavior and the parent role. Items are assessed on a 5- point Likert scale, from "Strongly disagree" (1) to "Strongly agree" (5).
Parent emotion regulation | immediately post first-stage intervention (4 weeks following baseline)
  The Parent Emotion Regulation Scale (PERS; Perreira, Barros, Roberto, & Marques, 2017) is a 20-item measure of parents' emotion regulation abilities. The PERS assesses four dimensions of parent emotion regulation (orientation to the child's emotions, avoidance of the child's emotions, lack of emotional control and acceptance of the child's and their own emotions), using a five-point Likert scale (from "Never or almost never" to "Always or almost always").
Changes in parent emotion regulation | post second-stage intervention (8 weeks following baseline)
  The Parent Emotion Regulation Scale (PERS; Perreira, Barros, Roberto, & Marques, 2017) is a 20-item measure of parents' emotion regulation abilities. The PERS assesses four dimensions of parent emotion regulation (orientation to the child's emotions, avoidance of the child's emotions, lack of emotional control and acceptance of the child's and their own emotions), using a five-point Likert scale (from "Never or almost never" to "Always or almost always").
Changes in parent emotion regulation - follow up | 6-month follow-up
  The Parent Emotion Regulation Scale (PERS; Perreira, Barros, Roberto, & Marques, 2017) is a 20-item measure of parents' emotion regulation abilities. The PERS assesses four dimensions of parent emotion regulation (orientation to the child's emotions, avoidance of the child's emotions, lack of emotional control and acceptance of the child's and their own emotions), using a five-point Likert scale (from "Never or almost never" to "Always or almost always").
Changes in parent emotion regulation - follow up one year | 12-month follow-up
  The Parent Emotion Regulation Scale (PERS; Perreira, Barros, Roberto, & Marques, 2017) is a 20-item measure of parents' emotion regulation abilities. The PERS assesses four dimensions of parent emotion regulation (orientation to the child's emotions, avoidance of the child's emotions, lack of emotional control and acceptance of the child's and their own emotions), using a five-point Likert scale (from "Never or almost never" to "Always or almost always").
Child attachment (moderator variable) | baseline
  The Security Scale (Kerns, Klepac, & Cole, 1996) is a 15-item measure of attachment security in children aged 8 to 12. The scale uses a "some kids... other kids..." format and asks respondents to select the degree to which they feel they are similar to the type of children they have previously selected, using a two-point Likert scale ("Really true for me" or "Sort of true for me".
Academic burnout | Baseline
  The School Burnout Inventory (Salmela-Aro et al., 2009) consists of 9 items that measure three aspects of school burnout, namely, exhaustion at school, cynicism toward the meaning of school, and the sense of inadequacy at school.
Changes in academic burnout | post second-stage intervention (8 weeks following baseline)
  The School Burnout Inventory (Salmela-Aro et al., 2009) consists of 9 items that measure three aspects of school burnout, namely, exhaustion at school, cynicism toward the meaning of school, and the sense of inadequacy at school.

CONTACTS AND LOCATIONS:
Locations (1):
- Oana David, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: No